CLINICAL TRIAL: NCT00517829
Title: Phase II Trial of Docetaxel Plus Oxaliplatin (DOCOX) With or Without Cetuximab in Patients With Metastatic Gastric and/or Gastroesophageal Junction Adenocarcinoma
Brief Title: Docetaxel+Oxali+/-Cetux Met Gastric/GEJ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Eli Lilly and Company (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06063
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Gastric Cancer Adenocarcinoma Metastatic
Keywords: metastatic gastric or adenocarcinoma of the GE junction
MeSH Terms: interventions — Docetaxel; Cetuximab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- Docetaxel plus Oxaliplatin (Active Comparator): Docetaxel as an intravenous (IV) infusion over 1 hour, followed by oxaliplatin IV over 2 hours
  Interventions: Drug: Docetaxel; Drug: oxaliplatin
- 2- Docetaxel plus oxaliplatin plus cetuximab (Active Comparator): Docetaxel 60 mg/m2 as an IV infusion over 1 ho ur, followed by oxaliplatin 130 mg/m2 IV over 2 hours, followed by cetuximab 400 mg/m2 IV over 120 minutes (first dose only), all other doses are 250 mg/m2 over 60 minutes.
  Interventions: Drug: Docetaxel; Drug: cetuximab; Drug: oxaliplatin

INTERVENTIONS:
Drug: Docetaxel — Taxotere 60 mg/m2 as an intravenous (IV) infusion over 1 hour
  Other Names: Taxotere (docetaxel)
Drug: cetuximab — ERBITUX 400 mg/m2 IV over 120 minutes (first dose only), all other doses are 250 mg/m2 over 60 minutes.
  Other Names: ERBITUX (cetuximab)
  Arms: 2- Docetaxel plus oxaliplatin plus cetuximab
Drug: oxaliplatin — Eloxatin 130 mg/m2 IV over 2 hours
  Other Names: Eloxatin (oxaliplatin)

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) docetaxel, oxaliplatin, and cetuximab have on gastric or GEJ cancer.

DETAILED DESCRIPTION:
This is a Phase II, open- label, randomized, noncomparative study. Patients will be stratified at randomization by ECOG PS. There is no intent to have equal numbers of patients for each PS (ie, 0, 1, and 2), but rather stratification will be conducted to ensure that the 2 treatment arms are well-balanced for ECOG PS.

Patients will be randomly assigned to either Arm 1 - Taxotere 60 mg/m2 as an intravenous (IV) infusion over 1 hour, followed by Eloxatin 130 mg/m2 IV over 2 hours or Arm 2 - Taxotere 60 mg/m2 as an IV infusion over 1 ho ur, followed by Eloxatin 130mg/m2 IV over 2 hours, followed by ERBITUX 400 mg/m2 IV over 120 minutes (first dose only), all other doses are 250 mg/m2 over 60 minutes. Taxotere and Eloxatin will be given on Day 1 of each 21-day cycle; ERBITUX is given on Days 1, 8, and 15 of each cycle.

Treatment will continue until disease progression or intolerable toxicity. Patients who achieve a CR will receive an additional 2 cycles of treatment. Patients will be limited to 24 months of participation, counted from the date of the first dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically confirmed Stage IV adenocarcinoma of the GEJ/stomach

Note: Adjuvant radiation plus treatment with 5-FU and leucovorin is permitted, but not required.

* Patients must have measurable disease
* Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2
* Patient is greater than 18 years of age
* If present, any pre-existing (current) peripheral neuropathy must be ≤ Grade 1
* Patient's laboratory values must fall within the limits set forth in section 4.2 of the protocol
* Patient has a negative serum pregnancy test within 7 days prior to registration (female patients of childbearing potential)
* If fertile, patient (male or female) has agreed to use an acceptable method of birth control to avoid pregnancy for the duration of the study and for a 2 month period thereafter
* Patient (or guardian) has signed a Patient Informed Consent Form
* Patient (or guardian) has signed a Patient Authorization Form

Exclusion Criteria:

* Patient has any metastatic disease other than that defined in section 4.2 (criterion #1)
* Patient has had prior treatment that included anything other than adjuvant radiation plus treatment with 5-FU and leucovorin. Prior treatment must have been completed > 6 months prior to registration in current study. No other prior regimens are allowed.

Note: Adjuvant radiation plus treatment with 5-FU and leucovorin is permitted, but not required.

* If present, any peripheral neuropathy is > Grade 1
* Patient has a known hypersensitivity to Taxotere (or any drug formulated with Polysorbate-80), or Eloxatin
* Has had a prior severe infusion reaction (Grade 4) to a monoclonal antibody
* Has received prior therapy, at any time, which specifically and directly targets the EGFR pathway
* Patient is receiving concurrent immunotherapy or any other concurrent treatment for their cancer
* Has had prior stem cell or bone marrow transplant or any organ transplant with the exception of corneal transplant or cadaver bone graft
* Has a significant history of uncontrolled cardiac disease; ie, uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, or cardiomyopathy with decreased ejection fraction (LVEF<50%)
* Has evidence of CNS involvement (CNS imaging is not required for study enrollment unless clinically suspected CNS disease is present.)
* Patient has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection
* Patient is known to be HIV positive or have a history of hepatitis B or C
* Patient has a history of other malignancy within the last 5 years (except for squamous or basal cell carcinoma of the skin, carcinoma in situ of the cervix , or superficial transitional cell carcinoma of the bladder), which could affect the diagnosis or assessment of current condition.
* Patient is a pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Richards, MD, Principal Investigator — US Oncology Research
Locations (46):
- United States (46):
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Rocky Mountain Cancer Center - Midtown, Denver, Colorado
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hope Center, Terre Haute, Indiana
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - New York Oncology Hematology, P.C., Hudson, New York
  - Interlakes Oncology Hematology, PC, Rochester, New York
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Mahoning Valley Hematology Oncology Associates, Boardman, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Texas Oncology, P.A. Amarillo, Amarillo, Texas
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, P.A. - Bedford, Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Methodist Charlton Cancer Ctr., Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Texas Oncology, P.A., Garland, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - Texas Oncology - Odessa, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer and Research, Waco, Texas
  - Fairfax Northern VA Hem-Onc PC, Arlington, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onc and Hem Associates of SW VA, Inc., Salem, Virginia
  - Puget Sound Cancer Center - Edmonds, Edmonds, Washington
  - Columbia Basin Hematology & Oncology, Kennewicke, Washington
  - Puget Sound Cancer Center - Seattle, Seattle, Washington
  - Cancer Care Northwest - South, Spokane, Washington
  - Northwest Cancer Specialist - Vancouver, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richards D, Kocs DM, Spira AI, David McCollum A, Diab S, Hecker LI, Cohn A, Zhan F, Asmar L. Results of docetaxel plus oxaliplatin (DOCOX) +/- cetuximab in patients with metastatic gastric and/or gastroesophageal junction adenocarcinoma: results of a randomised Phase 2 study. Eur J Cancer. 2013 Sep;49(13):2823-31. doi: 10.1016/j.ejca.2013.04.022. Epub 2013 Jun 5. PMID 23747051

RESULTS

PARTICIPANT FLOW:
Groups:
- DOCOX: Docetaxel 60 mg/m2 + Oxaliplatin 130 mg/m2 every 21 days
- DOCOX+Cebuximab: Docetaxel 60 mg/m2 + Oxaliplatin 130 mg/m2 + Cetuximab 400 mg/m2 (first dose only, subsequent doses 250 mg/m2) every 21 days
Period: Overall Study
Arm/Group | DOCOX | DOCOX+Cebuximab
Started | 75 | 75
Completed | 0 | 0
Not Completed | 75 | 75
Not completed — Adverse Event | 22 | 34
Not completed — Disease Progression | 39 | 32
Not completed — Patient Request | 6 | 5
Not completed — Investigator Request | 5 | 3
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | DOCOX | DOCOX+Cebuximab | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.9) | 61.5 (11.5) | 61.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 59 | 60 | 119
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 62 | 56 | 118
  Black | 5 | 7 | 12
  Hispanic | 5 | 9 | 14
  Asian | 3 | 1 | 4
  Hawaiian | 0 | 1 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: PFS is measured from the date of randomization to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Treatment will continue until disease progression or intolerable toxicity, up to 2 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DOCOX | DOCOX+Cebuximab
Number analyzed (Participants) | 75 | 75
months | 4.7 [3.0 to 5.6] | 5.1 [4.3 to 5.9]

2. Secondary Outcome: Overall Survival
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: Treatment will continue until disease progression or intolerable toxicity
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DOCOX | DOCOX+Cebuximab
Number analyzed (Participants) | 75 | 75
months | 8.5 [7.1 to 12.0] | 9.4 [6.7 to 10.1]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: Treatment will continue until disease progression or intolerable toxicity.
Population: Evaluable Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DOCOX | DOCOX+Cebuximab
Number analyzed (Participants) | 68 | 71
percentage of participants | 26.5 [16.5 to 38.6] | 38.0 [26.8 to 50.3]

4. Secondary Outcome: Time to Response
Description: For patients who achieve a major objective response (CR or PR) the time to response will be assessed as the date of registration to the date of response.
Time Frame: Treatment will continue until disease progression or intolerable toxicity
Population: Patients who achieve a major objective response (CR or PR)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DOCOX | DOCOX+Cebuximab
Number analyzed (Participants) | 18 | 27
months | 1.3 [1.1 to 5.2] | 1.4 [1.1 to 4.0]

5. Secondary Outcome: Duration of Response
Description: The duration of response is measured from the time measurement criteria are first met for CR/PR until the first date that recurrent or progressive disease is objectively documented.
Time Frame: Treatment will continue until disease progression or intolerable toxicity
Population: Patients who achieve a major objective response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DOCOX | DOCOX+Cebuximab
Number analyzed (Participants) | 18 | 27
months | 7.3 [1.5 to 23.7] | 5.6 [2.3 to 13.2]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | DOCOX | DOCOX+Cebuximab
Serious Adverse Events (participants affected / at risk) | 20/68 | 26/72
Other Adverse Events (participants affected / at risk) | 65/68 | 67/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOCOX (N=68) | DOCOX+Cebuximab (N=72)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CACHEXIA (Investigations) | 0 (0) | 1 (1)
CANCER (Investigations) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 1 (1)
CHOLANGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 2 (3)
DEFICIENCY VITAMIN (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 4 (4) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 5 (5) | 4 (6)
EDEMA LARYNX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EDEMA SCROTAL (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ESOPHAGEAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 1 (1)
FEBRILE NEUTROPENIA (Infections and infestations) | 7 (7) | 13 (14)
FEVER (General disorders) | 1 (1) | 1 (1)
FIBRILLATION ATRIAL (Cardiac disorders) | 0 (0) | 1 (1)
GASTRIC ULCER PERFORATED (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 2 (2) | 0 (0)
HYPERSENSITIVITY REACTION (NOS) (Nervous system disorders) | 0 (0) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOXEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
IMBALANCE BLOOD ELECTROLYTE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 2 (3) | 1 (1)
INFECTION BLADDER (Renal and urinary disorders) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LUNG FIBROSIS INTERSTITIAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NEUROPATHY (Nervous system disorders) | 0 (0) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
PERFORATION GASTROINTESTINAL (Gastrointestinal disorders) | 0 (0) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SHOCK (Nervous system disorders) | 1 (1) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
SWEATING (General disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (2)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
WEAKNESS GENERALIZED (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOCOX (N=68) | DOCOX+Cebuximab (N=72)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 5 (6)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 6 (6)
ALOPECIA (Skin and subcutaneous tissue disorders) | 22 (24) | 17 (19)
ANEMIA (Blood and lymphatic system disorders) | 19 (43) | 19 (31)
ANOREXIA (Gastrointestinal disorders) | 13 (28) | 12 (16)
CONSTIPATION (Gastrointestinal disorders) | 10 (11) | 13 (19)
DEHYDRATION (Gastrointestinal disorders) | 9 (13) | 11 (20)
DIARRHEA (Gastrointestinal disorders) | 26 (39) | 34 (92)
DIZZINESS (Nervous system disorders) | 1 (1) | 6 (6)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (10)
FATIGUE (General disorders) | 33 (75) | 36 (81)
FEVER (Gastrointestinal disorders) | 5 (6) | 2 (4)
FLUSHING (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
HEADACHE (General disorders) | 4 (4) | 4 (4)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (6) | 5 (12)
HYPERSENSITIVITY REACTION (NOS) (Nervous system disorders) | 3 (3) | 9 (12)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (4) | 4 (10)
HYPOKALEMIA (Metabolism and nutrition disorders) | 5 (5) | 5 (10)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 4 (4) | 14 (39)
INSOMNIA (General disorders) | 1 (1) | 4 (7)
IRRITATION SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
LEUKOPENIA (Blood and lymphatic system disorders) | 13 (26) | 14 (47)
MUCOSITIS ORAL (Gastrointestinal disorders) | 3 (4) | 8 (11)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (8)
NAUSEA (Gastrointestinal disorders) | 26 (37) | 27 (53)
NEUROPATHY (Nervous system disorders) | 17 (23) | 9 (14)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 12 (18) | 16 (34)
NEUTROPENIA (Blood and lymphatic system disorders) | 45 (141) | 41 (119)
PAIN (General disorders) | 3 (3) | 7 (8)
PAIN MOUTH (Gastrointestinal disorders) | 1 (1) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 2 (3) | 17 (36)
RASH ACNEFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 32 (58)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 8 (13)
TASTE ALTERATION (Gastrointestinal disorders) | 10 (13) | 8 (10)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 12 (41) | 8 (23)
TINGLING (Nervous system disorders) | 4 (11) | 4 (4)
VOMITING (Gastrointestinal disorders) | 14 (18) | 12 (20)
WEAKNESS GENERALIZED (General disorders) | 8 (11) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No